CLINICAL TRIAL: NCT04025476
Title: Clinical Observational Research on Changes of Peripheral Blood Mononuclear Cell（PBMC） Immunity and Expression Profile in Peripheral Blood of Different Course of of Vogt-Hoyanagi-Harada（VKH） Patients.
Brief Title: Immune Profile of Acute VKH Patients PBMC
Acronym: IPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: AFM1713D1
Record Dates: First submitted 2019-07-14; First posted 2019-07-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: VKH Syndrome
Keywords: VKH; immune profile;
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome | interventions — Steroids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample of VKH patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VKH patients: acute VKH patients
  Interventions: Drug: Steroids
- control: health people age/sex match to the VKH patients

INTERVENTIONS:
Drug: Steroids — IV and oral steroids
  Groups: VKH patients

SUMMARY:
The investigators will collect blood samples of different courses of VKH patients for investigating immune profile, observe major immune cells number ,functional and membrane molecular changes in the course of treatment, to investigate pathogenesis of VKH. Meanwhile, the investigators will collect clinical data of VKH patients to observe choroid and retina change in different courses.

ELIGIBILITY:
Inclusion Criteria:

1. Acute VKH patients, meet a criterion of VKH, no recurrence.
2. Age range from 18 to 50 years old.

Exclusion Criteria:

1. Patients with Severe Cardiovascular and Cerebrovascular Diseases
2. Patients allergic to steroid or contrast agents;
3. A history of ocular trauma or intraocular surgery within 3 months; Vaccinated; History of infectious diseases
4. having a history of heredity, immune system correlation, neuroendocrine and digestive system diseases
5. Patients who take health care products for a long time and have heavy alcohol and tobacco addiction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: acute primary VKH patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-07 (Estimated)

PRIMARY OUTCOMES:
T/B /NK(natural killer )/monocyte...etc, cell numbers of blood samples in VKH patients | one year
  use flow cytometry to count T/B /NK/monocyte...etc, cell numbers
T/B /NK/monocyte...etc cell subtype proportion in blood samples in VKH patients | one year
  use flow cytometry to measure T/B /NK/monocyte...etc cell subtype proportion
T/B /NK/monocyte...etc cell functional change in VKH patients | one year
  use ELISA(enzyme linked immunosorbent assay) to measure inflammatory cytokines level in peripheral blood

SECONDARY OUTCOMES:
choroid and retinal thickness change in different course of VKH patients | one year
  Use OCT（optical coherence tomography） to measure choroid and retina thickness changes in macular zone of different course VKH patients
Use OCTA(optical coherence tomography angiography) to measure macular and optic disc vascular index | one year
  Use OCTA to measure macular and optic disc vascular index in different course VKH patients
Use Maia perimeter to measure macular integrality | one year
  Use Maia perimeter to measure macular integrality including light threshold and central fixation.
measure the Injury degree of choroid and retinal vessels | one year
  Use FFA(fluorescein fundus angiography)/ICG(Indocyanine Green Angiography) to measure the Injury degree of choroid and retinal vessels

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, MD, Study Director — Central-southern university, Aier ophthalmology colleage
Locations (1):
- Wuhan Aier eye hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No